CLINICAL TRIAL: NCT03201809
Title: Comparison of Preoperative Ultrasound Guided Pectoralis Nerve Block Placement Versus Intra-operative Placement: A Prospective Randomized Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 918749
Record Dates: First submitted 2017-06-21; First posted 2017-06-28 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two groups, conventional treatment versus experimental treatment; blocked randomization scheme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- On-Q Catheter (Experimental): On-Q catheters placed within the implant pocket; infusion of 0.2% Ropivacaine at 4 mL/h for a total of 400 mL (about 4 days).
  Interventions: Device: On-Q
- Ultrasound Guided Pectoral Nerve Block (Active Comparator): Single Shot Pre-operative injections of 10 mL of 0.25% Ropivicaine for the Pecs 1 injection, and 20 mL of 0.25% Ropivacaine for the pecs 2 injection
  Interventions: Drug: Ultrasound guided pectoral nerve block

INTERVENTIONS:
Device: On-Q — 0.2% Ropivicaine at 4 mL/h via On-Q catheter placed sub-pectoral
  Arms: On-Q Catheter
Drug: Ultrasound guided pectoral nerve block — Single Shot Pre-operative injections of 10 mL of 0.25% Ropivicaine for the Pecs 1 injection, and 20 mL of 0.25% Ropivacaine for the Pecs 2 injection
  Arms: Ultrasound Guided Pectoral Nerve Block

SUMMARY:
This study investigates the use of post-operative on-Q pain catheters for tissue expander based breast reconstruction, versus conventional ultrasound-guided blocks placed pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

* presenting for breast reconstruction w/ planned two-stage, sub muscular tissue expander placement.

Exclusion Criteria:

* pregnant, prisoners, cannot consent, history of chronic pain or pain medication use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Wong, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
available only as aggregate / HIPAA non-identifiable data in published papers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | On-Q Catheter | Ultrasound Guided Pectoral Nerve Block
Started | 6 | 6
Completed | 4 | 6
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On-Q Catheter | Ultrasound Guided Pectoral Nerve Block | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 42.8 [41 to 64] | 50.7 [33 to 63] | 48.1 [33 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Narcotic Usage
Description: amount of narcotic used
Time Frame: post operation up to 2 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | On-Q Catheter | Ultrasound Guided Pectoral Nerve Block
Number analyzed (Participants) | 6 | 6
mg | 23.95 (24.32) | 6.43 (5.95)

2. Secondary Outcome: Post-operative Anti-emetic Usage
Description: number and amount of anti-emetic used
Time Frame: post operation up to 2 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | On-Q Catheter | Ultrasound Guided Pectoral Nerve Block
Number analyzed (Participants) | 6 | 6
mg | 3.11 (3.33) | 2.00 (2.31)

3. Secondary Outcome: Post-operative Self-reported Pain Scores
Description: Pain scores overall and by breast: 0 (no pain) - 100 (extreme pain) analog scale.
Time Frame: post operation up to 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | On-Q Catheter | Ultrasound Guided Pectoral Nerve Block
Number analyzed (Participants) | 6 | 6
score on a scale
  Pain Level in Breasts Overall at Rest (Postop 7 days) | 20.50 (19.09) | 24.33 (12.66)
  Pain Level in Breasts Overall with Activity (Postop 7 days) | 38.00 (33.94) | 56.33 (19.43)
  Pain Level in Left Breast at Rest (Postop 7 days) | 36.00 (36.77) | 17.00 (4.36)
  Pain Level in Left Breast with Activity (Postop 7 days) | 37.00 (31.11) | 31.67 (15.04)
  Pain Level in Right Breast at Rest (Postop 7 days): | 24.50 (21.92) | 30.67 (17.67)
  Pain Level in Right Breast with Activity (Postop 7 days) | 32.50 (26.16) | 56.00 (20.30)

ADVERSE EVENTS:
Time Frame: Up to 10 days
Arm/Group | On-Q Catheter | Ultrasound Guided Pectoral Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Due to 2 patients being lost to follow up and the small total number of subjects, the study findings were limited. Because of the nominal number of breast reconstruction patients at our institution meeting inclusion criteria for this trial, there was low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT03201809/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT03201809/ICF_001.pdf